CLINICAL TRIAL: NCT02013544
Title: Intravaginal Prasterone (DHEA) Against Vulvovaginal Atrophy Associated With Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EndoCeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-238
Record Dates: First submitted 2013-12-09; First posted 2013-12-17 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Vaginal Atrophy
Keywords: Vulvovaginal atrophy (VVA); Vaginal atrophy; Atrophic vaginitis; prasterone; DHEA; Intrarosa
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo vaginal ovule daily for 12 weeks
  Interventions: Drug: Placebo
- Prasterone (Experimental): Prasterone (DHEA) vaginal ovule daily for 12 weeks
  Interventions: Drug: Prasterone (DHEA)

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Prasterone (DHEA)
  Arms: Prasterone

SUMMARY:
The purpose of this study is to confirm the efficacy of intravaginal prasterone (DHEA) on symptoms of vulvovaginal atrophy due to menopause and to collect further data on subjects exposed to intravaginal DHEA in order to meet the ICH E1 guideline requirements.

ELIGIBILITY:
Inclusion Criteria:

Main criteria:

* Postmenopausal women (hysterectomized or not)
* Women between 40 and 80 years of age
* Women having ≤5% of superficial cells on vaginal smear at baseline
* Women having a vaginal pH above 5 at baseline
* Women who have self-identified moderate or severe symptom(s) of vaginal atrophy
* Willing to participate in the study and sign an informed consent

Exclusion Criteria:

Main criteria:

* Previous enrollment in EndoCeutics studies performed with intravaginal DHEA
* Previous diagnosis of cancer, except skin cancer (non melanoma)
* Clinically significant metabolic or endocrine disease (including diabetes mellitus) not controlled by medication
* The administration of any investigational drug within 30 days of screening visit
* Clinically significant abnormal serum biochemistry, urinalysis or hematology

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernand Labrie, M.D., Ph.D., Study Chair — EndoCeutics Inc.; David F Archer, M.D., Principal Investigator — Clinical Research Center, Eastern Virginia Medical School, Norfolk, VA
Locations (38):
- United States (24):
  - EndoCeutics site # 39, Montgomery, Alabama
  - EndoCeutics site # 14, Tucson, Arizona
  - EndoCeutics site # 21, Sacramento, California
  - EndoCeutics site # 83, San Diego, California
  - EndoCeutics site # 30, San Diego, California
  - EndoCeutics site # 36, Denver, Colorado
  - EndoCeutics site # 52, Denver, Colorado
  - EndoCeutics site # 45, Boynton Beach, Florida
  - EndoCeutics site # 60, Lake Worth, Florida
  - EndoCeutics site # 54, North Miami, Florida
  - EndoCeutics site # 80, West Palm Beach, Florida
  - EndoCeutics site # 23, Atlanta, Georgia
  - EndoCeutics site # 55, Wichita, Kansas
  - EndoCeutics site # 86, Louisville, Kentucky
  - EndoCeutics site # 27, Lutherville, Maryland
  - EndoCeutics site # 87, Lawrenceville, New Jersey
  - EndoCeutics site # 81, Plainsboro, New Jersey
  - EndoCeutics site # 05, Cleveland, Ohio
  - EndoCeutics site # 15, Columbus, Ohio
  - EndoCeutics site # 75, Philadelphia, Pennsylvania
  - EndoCeutics site # 84, Corpus Christi, Texas
  - EndoCeutics site # 82, Houston, Texas
  - EndoCeutics site # 03, Norfolk, Virginia
  - EndoCeutics site # 76, Seattle, Washington
- Canada (14):
  - EndoCeutics site # 85, Burlington, Ontario
  - EndoCeutics site # 69, Corunna, Ontario
  - EndoCeutics site # 68, Sarnia, Ontario
  - EndoCeutics site # 73, Waterloo, Ontario
  - EndoCeutics site # 04, Drummondville, Quebec
  - EndoCeutics site # 12, Montreal, Quebec
  - EndoCeutics site # 79, Pointe-Claire, Quebec
  - EndoCeutics site # 02, Québec, Quebec
  - EndoCeutics site # 01, Québec, Quebec
  - EndoCeutics site # 77, Québec, Quebec
  - EndoCeutics site # 78, Québec, Quebec
  - EndoCeutics site # 18, Saint Romuald, Quebec
  - EndoCeutics site # 74, Sherbrooke, Quebec
  - EndoCeutics site # 67, Victoriaville, Quebec

REFERENCES:
- [Result] Ke Y, Labrie F, Gonthier R, Simard JN, Bergeron D, Martel C, Vaillancourt M, Montesino M, Lavoie L, Archer DF, Balser J, Moyneur E; other participating Members of the Prasterone Clinical Research Group. Serum levels of sex steroids and metabolites following 12 weeks of intravaginal 0.50% DHEA administration. J Steroid Biochem Mol Biol. 2015 Nov;154:186-96. doi: 10.1016/j.jsbmb.2015.08.016. Epub 2015 Aug 17. PMID 26291918
- [Result] Labrie F, Derogatis L, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; Members of the VVA Prasterone Research Group. Effect of Intravaginal Prasterone on Sexual Dysfunction in Postmenopausal Women with Vulvovaginal Atrophy. J Sex Med. 2015 Dec;12(12):2401-12. doi: 10.1111/jsm.13045. Epub 2015 Nov 23. PMID 26597311
- [Result] Labrie F, Montesino M, Archer DF, Lavoie L, Beauregard A, Cote I, Martel C, Vaillancourt M, Balser J, Moyneur E; other participating Members of the Prasterone Clinical Research Group. Influence of treatment of vulvovaginal atrophy with intravaginal prasterone on the male partner. Climacteric. 2015;18(6):817-25. doi: 10.3109/13697137.2015.1077508. Epub 2015 Oct 30. PMID 26517756
- [Result] Labrie F, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Research Group. Efficacy of intravaginal dehydroepiandrosterone (DHEA) on moderate to severe dyspareunia and vaginal dryness, symptoms of vulvovaginal atrophy, and of the genitourinary syndrome of menopause. Menopause. 2016 Mar;23(3):243-56. doi: 10.1097/GME.0000000000000571. PMID 26731686
- [Result] Martel C, Labrie F, Archer DF, Ke Y, Gonthier R, Simard JN, Lavoie L, Vaillancourt M, Montesino M, Balser J, Moyneur E; other participating members of the Prasterone Clinical Research Group. Serum steroid concentrations remain within normal postmenopausal values in women receiving daily 6.5mg intravaginal prasterone for 12 weeks. J Steroid Biochem Mol Biol. 2016 May;159:142-53. doi: 10.1016/j.jsbmb.2016.03.016. Epub 2016 Mar 10. PMID 26972555
- [Result] Montesino M, Labrie F, Archer DF, Zerhouni J, Cote I, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Moyneur E, Balser J. Evaluation of the acceptability of intravaginal prasterone ovule administration using an applicator. Gynecol Endocrinol. 2016;32(3):240-5. doi: 10.3109/09513590.2015.1110140. Epub 2016 Jan 6. PMID 26634942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1226 subjects were screened at 38 medical/research sites located in the US (24 centers) and Canada (14 centers) and 558 subjects were randomized. The first subject first visit was on 11-FEB-2014 and the last subject last visit was on 06-JAN-2015.
Groups:
- Placebo: Placebo: Placebo vaginal ovule; daily dosing with one ovule for 12 weeks
- 0.50% Prasterone (DHEA): Prasterone (DHEA): Vaginal ovule containing 0.50% (6.5 mg) prasterone; daily dosing with one ovule for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Started | 182 | 376
Safety Population | 180 | 374
ITT Population | 157 | 325
Completed | 171 | 356
Not Completed | 11 | 20
Not completed — Adverse Event | 5 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Physician Decision | 0 | 1
Not completed — Entry criteria not met/non-compliance | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population corresponds to the Safety Population which includes all subjects who received any amount of prasterone or placebo, and who have any safety information available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.50% Prasterone (DHEA) | Total
Number analyzed (Participants) | 180 | 374 | 554
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.55 (5.75) | 59.51 (6.78) | 59.53 (6.46)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 180 | 374 | 554
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Caucasian | 163 | 338 | 501
  Black or African American | 13 | 28 | 41
  Asian | 2 | 4 | 6
  American Indian or Alaska Native | 0 | 1 | 1
  Native hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Percentage of Superficial Cells in the Maturation Index of the Vaginal Smear
Description: The percentage of superficial cells was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: Efficacy analyses were performed primarily on the Intent to Treat (ITT) population defined as all subjects who have received at least one dose of study drug with a baseline (Day 1) evaluation meeting the study entry criteria.
Measure: Mean (Standard Error); unit: Percentage of superficial cells
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 157 | 325
Percentage of superficial cells
  Baseline | 1.04 (0.11) | 1.02 (0.08)
  Week 12 | 2.78 (0.27) | 11.22 (0.56)
  Change from Baseline to Week 12 | 1.75 (0.27) | 10.20 (0.57)

2. Primary Outcome: Change From Baseline to Week 12 in Percentage of Parabasal Cells in the Maturation Index of the Vaginal Smear
Description: The percentage of parabasal cells was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage of parabasal cells
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 157 | 325
Percentage of parabasal cells
  Baseline | 51.66 (3.00) | 54.25 (2.14)
  Week 12 | 39.68 (2.68) | 12.74 (1.02)
  Change from Baseline to Week 12 | -11.98 (2.36) | -41.51 (2.01)

3. Primary Outcome: Change From Baseline to Week 12 in Vaginal pH
Description: A pH strip fixed on an Ayre spatula (or equivalent) was applied directly to the lateral wall of the vagina. The change in color of the pH indicator strip was compared to the color chart for pH evaluation. The corresponding pH value (with one decimal) was recorded. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 157 | 325
units on a scale
  Baseline | 6.32 (0.05) | 6.34 (0.04)
  Week 12 | 6.05 (0.07) | 5.39 (0.05)
  Change from Baseline to Week 12 | -0.27 (0.06) | -0.94 (0.05)

4. Primary Outcome: Change From Baseline to Week 12 in Severity of the Most Bothersome Symptom of Dyspareunia
Description: The severity of dyspareunia was evaluated by a questionnaire filled out by women. The severity of dyspareunia recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 157 | 325
units on a scale
  Baseline | 2.56 (0.04) | 2.54 (0.03)
  Week 12 | 1.50 (0.08) | 1.13 (0.05)
  Change from Baseline to Week 12 | -1.06 (0.08) | -1.42 (0.06)

5. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Dryness
Description: The severity of vaginal dryness was evaluated by a questionnaire filled out by women. The severity of vaginal dryness recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: Efficacy analyses on vaginal dryness were performed on a sub-group of the Intent to Treat (ITT) population (defined as all subjects who have received at least one dose of study drug with a baseline (Day 1) evaluation meeting the study entry criteria) who had self-identified moderate to severe vaginal dryness at Baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 132 | 273
units on a scale
  Baseline | 2.30 (0.04) | 2.30 (0.03)
  Week 12 | 1.13 (0.08) | 0.86 (0.05)
  Change from Baseline to Week 12 | -1.17 (0.09) | -1.44 (0.06)

6. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Secretions
Description: To evaluate the aspect of the mucosa and the local tolerance to prasterone ovules, the vaginal secretions (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy were analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 157 | 325
units on a scale
  Baseline | 2.63 (0.05) | 2.70 (0.04)
  Week 12 | 2.24 (0.06) | 1.97 (0.04)
  Change from Baseline to Week 12 | -0.39 (0.06) | -0.73 (0.04)

7. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Epithelial Integrity
Description: To evaluate the aspect of the mucosa and the local tolerance to prasterone ovules, the vaginal epithelial integrity (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 157 | 325
units on a scale
  Baseline | 2.43 (0.06) | 2.45 (0.05)
  Week 12 | 2.06 (0.06) | 1.75 (0.04)
  Change from Baseline to Week 12 | -0.37 (0.07) | -0.69 (0.05)

8. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Epithelial Surface Thickness
Description: To evaluate the aspect of the mucosa and the local tolerance to prasterone ovules, the vaginal epithelial surface thickness (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 157 | 325
units on a scale
  Baseline | 2.76 (0.05) | 2.83 (0.03)
  Week 12 | 2.41 (0.05) | 2.09 (0.04)
  Change from Baseline to Week 12 | -0.36 (0.06) | -0.74 (0.05)

9. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Color
Description: To evaluate the aspect of the mucosa and the local tolerance to prasterone ovules, the vaginal color (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Number analyzed (Participants) | 157 | 325
units on a scale
  Baseline | 2.67 (0.05) | 2.75 (0.03)
  Week 12 | 2.34 (0.05) | 2.03 (0.04)
  Change from Baseline to Week 12 | -0.33 (0.06) | -0.73 (0.05)

ADVERSE EVENTS:
Time Frame: From Baseline to Week 12 (+ 30-day follow-up period after last dose)
Arm/Group | Placebo | 0.50% Prasterone (DHEA)
Serious Adverse Events (participants affected / at risk) | 0/180 | 5/374
Other Adverse Events (participants affected / at risk) | 10/180 | 24/374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=180) | 0.50% Prasterone (DHEA) (N=374)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Post-procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastric bypass (Surgical and medical procedures) | 0 | 1
Hernia hiatus repair (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=180) | 0.50% Prasterone (DHEA) (N=374)
Application site discharge (General disorders) | 10 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall provide to the SPONSOR 30 days prior to submission all documents for publication, presentation, etc that report any trial results. The SPONSOR shall have editorial rights on documents and the right to review/comment with regard to (1) proprietary information, (2) accuracy of the information, (3) correctness of the scientific evaluation/conclusions and (4) to ensure that the information is fairly balanced and in compliance with regulations.